CLINICAL TRIAL: NCT03729843
Title: Cone Beam Computed Tomography Versus Intraoral Digital Radiography in Detection and Measurements of Simulated Periodontal Bone Defects Diagnostic Accuracy Study
Brief Title: Cone Beam Computed Tomography Versus Intraoral Digital Radiography in Detection and Measurements of Simulated Periodontal Bone Defects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marwa Mohamed Ali (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Ali, Lecturer Assistant of Oral Radiology Department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: HPHH
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Periodontal Bone Defects Will be Detected and Measured by 2 Techniques CBCT and Intraoral Digital Radiography to Compare the Accuracy of These Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT and intraoral digital radiography: simulated bone defects will be detected and measured by 2 techniques using CBCT and using intraoral digital radiography and the all measurements will be compared with the gold standard real measurements on the dry jaws
  Interventions: Radiation: CBCT and intraoral digital radiography

INTERVENTIONS:
Radiation: CBCT and intraoral digital radiography — Simulated periodontal bone defects will be measured by 2 techniques: group I detected and measured using CBCT and group II intraoral digital radiography and all the measurements will be compared with the gold standard real measurements on the dry jaws

SUMMARY:
The selection of a regenerative approach is primarily based on the configuration of the intrabony defect and esthetic risk of treatment. Accurate diagnosis of periodontal bone defects, such as vertical bone defects or furcation involvements, is a challenge for dental clinicians. A deficiency in comprehensive diagnosis may result in: 1) compromised prognosis of teeth; 2) changes in treatment plan; 3) unnecessary treatment; 4) longer treatment time; and 5) unanticipated treatment costs.

Thus, it is very important to have access to accurate diagnostic tools that can aid clinicians in cultivating an appropriate treatment choice. Periodontal assessments utilizing both clinical and radiographic examinations allow for the establishment of an accurate diagnosis as well as subsequent treatment choices.

Radiography plays an important role in periodontal diagnosis mainly because radiographs can reveal the amount and type of damage caused to the alveolar bone.

Digital imaging technique has created challenging opportunities for dental radiographic diagnosis. Digora was the first digital system for dental radiography based on a photostimulable phosphor technology.

E9ickholz et al. at 1999 compared linear measurements of interproximal bone loss on digitized radiographic images after application of different filters to the gold standard of intrasurgical measurements they concluded that all radiographic assessments on the digitized images came close to the intasurgical gold standard.

2D technologies do not allow for measurement of the bucco-lingual (B-L) width of the defect. Only the vertical height and the mesio-distal (M-D) width of the defect can be measured with 2D images.

Use of 3D volumetric images and 2D images in artificial bone defects have shown that CBCT has a sensitivity of 80% to 100% in detection and classification of bone defects, while intraoral radiographs present a sensitivity of 63% to 67%.

When compared with periapical and panoramic images, the CBCT has also shown an absence of distortion and overlapping, and the dimensions of the images that it presents were compatible with the actual size of the individual.

A few studies have been published comparing CBCT with digital radiography for the detection and measurements of periodontal bone defects.

DETAILED DESCRIPTION:
Periodontal disease is caused by an imbalance between bone formation and resorption, leading to an ultimate reduction in bone height. Detection of periodontal disease is important in the prevention of tooth loss. The detection and accurate assessment of the location, extent and configuration of the endosseous defect is important for the determination of the tooth prognosis, the treatment plan and the maintenance procedures.

Regenerative therapies for both intrabony and furcation defects are viable options, but early management of these defects offers the greatest potential for periodontal health. Intrabony defect morphology as well as degree of furcation involvement may affect overall regenerative outcomes and/or optimal treatment strategies.

Radiographic bone loss is also useful for assigning descriptors to indicate severity of periodontitis: <1/3 bone loss = mild, 1/3 to ½ bone loss = moderate, and >½ bone loss = severe. Classification of bony defects given by Papapanou et al. 2000 was used to differentiate bone defects into: Suprabony defects (SB), Infrabony defects (IB), Interradicular defects (IR).For classifying the intrabony defects (IT), the investigators used classification system by Goldman and Cohen 1958 which classified the IT defects into: 1 wall, 2 wall , 3 wall and Combined bone defects (CB). Other bone defects (OB) were classified by their topography as:Bulbous bone contour (BB), Reversed architecture (RA), Dehiscence (DH).

The potentially existing radiological furcation involvement was examined by identifying the furcation upper boundary and furcation lower boundary and was classified as Subclass A, B, and C according to the classification system by Tarnow and Fletcher 1984, where he added the vertical component to the diagnosis of furcation involvement. Subclass based on the vertical bone resorption from the furcation fornix was added.

* Subclass A: Denotes furcation involvements with vertical bone loss of 3 mm or less.
* Subclass B: Denotes furcation involvements with vertical bone loss from 4 to 6 mm.
* Subclass C: Presents with bone loss from the fornix of 7 mm or more.

  * The SB, IB, and OB defects were considered as absolute defects while IR defects were considered as relative defects because IR defects do not depict a particular bone lesion or defect rather they represent the stage in progress of periodontitis, i.e., once the periodontal disease progresses or its severity increases, it is bound to erode the bone between the multirooted teeth and involve the furcation.

Digital radiography is changing the diagnosis and treatment of dental diseases by incorporating computer technology into the field of dentistry. digital radiography have several advantages over film radiography, including immediate image production with solid-state devices; interactive display on a monitor with the ability to enhance image features and make direct linear and densitometric measurements; integrated storage; fast communication of images; lower contamination of the environment; security mechanisms to identify original images; ability to tag information such as a patient identifier, date of exposure and other relevant details; interoperability of the Digital Imaging and Communications in Medicine (DICOM) file format, which enables practitioners with different equipment and software to view and enhance the same images.

Furthermore, digital radiography offers a plethora of technical innovations to dentistry and is sure to significantly influence the arts of diagnosis, monitoring, research, as well as the treatment of dental diseases.

Cone beam computed tomography (CBCT) is a relatively new extra-oral imaging system which was specifically developed to overcome the limitations of periapical radiographs as it produces undistorted 3D information of the maxillofacial skeleton with a substantially lower radiation dose compared to conventional CT.

Consequently, CBCT has the potential to become non-invasive diagnostic instrument for various dental applications in which defect characterization, localization and volume measurements are important.

CBCT is currently being considered as a superior diagnostic tool for applications in periodontology. CBCT scanning was found to be more effective than other 2D imaging modalities in assessing periodontal structures. As CBCT had better potential of detecting periodontal bone defects in all directions compared with periapical radiographs. More over interproximal areas also, buccal and lingual defects could not be recognized from each other with intraoral radiographs.

ELIGIBILITY:
Inclusion Criteria:

* • The selected dry jaws should be intact with no mechanical damage (chips, cracks, or fractures in the alveolar process).

  * The teeth will be naturally attached to human jaws.
  * The study samples will not identified by age or gender group.

Exclusion Criteria:

* • teeth with metallic restorations to avoid artifacts generation on CBCT scanning.

  * Teeth with anomalies and fractures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patially or fully dentate dry jaws that match with the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2019-11-10 (Estimated); Study Completion 2020-11-10 (Estimated)

PRIMARY OUTCOMES:
CBCT and Intraoral Digital Radiography | 24 months
  Detection and measuring of artificially prepared periodontal bone defects.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Kandil, Professor, Study Chair — Cairo University